CLINICAL TRIAL: NCT03511131
Title: A Pragmatic Trial of An Adaptive eHealth HIV Prevention Program for Diverse Adolescent MSM
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Brian Mustanski, Professor, Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 5U01MD011281 (NIH); 5U01MD011281 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-27 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Hiv; Adolescent Behavior; Sex, Safe
Keywords: HIV prevention; Adolescent risk-taking behaviors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Adolescent Behavior; Safe Sex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- QSE Resp (Only follow) (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who responded to QSE, were randomized at month-6 to no additional treatment, and then followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed
- QSE Resp (KIU at 6-month) (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who responded to QSE, were randomized at month-6 to receive Keep It Up (KIU), and then followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up
- QSE Non-Resp, KIU-Control Resp (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who did not respond to QSE, were randomized at month-3 to receive Keep It Up-Control (KIU-Control), responded to KIU-Control at month-6, and then were followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up-Control
- QSE Non-Resp, KIU-Control Non-Resp, KIU (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who did not respond to QSE, were randomized at month-3 to receive Keep It Up-Control (KIU-Control), did not respond to KIU-Control at month-6, and so were randomized into Keep It Up (KIU). After KIU, they were followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up; Behavioral: Keep It Up-Control
- QSE Non-Resp, KIU Control Non-Resp, YMHP (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who did not respond to QSE, were randomized at month-3 to receive Keep It Up-Control (KIU-Control), did not respond to KIU-Control at month-6, and so were randomized into Young Men's Health Project (YMHP). After YMHP, they were followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up-Control; Behavioral: Young Men's Health Project
- QSE Non-Resp, KIU Resp (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who did not respond to QSE, were randomized at month-3 to receive Keep It Up (KIU), responded to KIU at month-6, and then were followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up
- QSE Non-Resp, KIU Non-Resp (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who did not respond to QSE, were randomized at month-3 to receive Keep It Up (KIU), did not respond to KIU at month-6, and then were randomized into no treatment/just follow for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up
- QSE Non-Resp, KIU Non-Resp, YMHP (Other): All participants enter Queer Sex Ed (QSE) and are measured at 0, 3, 6, 9, and 12-months. This arm is comprised of participants who did not respond to QSE, were randomized at month-3 to receive Keep It Up (KIU), did not respond to KIU at month-6, and then were randomized into Young Men's Health Project. After YMHP, they were followed for the rest of the study.
  Interventions: Behavioral: Queer Sex Ed; Behavioral: Keep It Up; Behavioral: Young Men's Health Project

INTERVENTIONS:
Behavioral: Queer Sex Ed — Comprehensive sexual health education program condition (Informational)
  Other Names: QSE, SMART Sex Ed
Behavioral: Keep It Up — Culturally/situation-relevant HIV-prevention experimental condition (Motivational/behavioral)
  Other Names: KIU, SMART Squad
  Arms: QSE Non-Resp, KIU Non-Resp; QSE Non-Resp, KIU Non-Resp, YMHP; QSE Non-Resp, KIU Resp; QSE Non-Resp, KIU-Control Non-Resp, KIU; QSE Resp (KIU at 6-month)
Behavioral: Keep It Up-Control — HIV knowledge control condition, attention-matched to KIU (Informational)
  Other Names: KIU-Control, SMART Sex Ed 2.0
  Arms: QSE Non-Resp, KIU Control Non-Resp, YMHP; QSE Non-Resp, KIU-Control Non-Resp, KIU; QSE Non-Resp, KIU-Control Resp
Behavioral: Young Men's Health Project — Motivational enhancement video interviewing condition (Motivational/behavioral)
  Other Names: YMHP, SMART Sessions
  Arms: QSE Non-Resp, KIU Control Non-Resp, YMHP; QSE Non-Resp, KIU Non-Resp, YMHP

SUMMARY:
This pragmatic trial of an HIV prevention program focuses on HIV risk-reduction in men who have sex with men (MSM) ages 13-18. The design is a three-tiered, internet-based HIV prevention intervention series that uses a sequential multiple assignment randomized trial (SMART) to track adolescent MSM reporting varying degree of sexual risk.The program package includes: (1-low risk) a universally-delivered, brief, online sexual health education program designed for sexual and gender minority youth regardless of whether they are sexually active (Queer Sex Ed); (2-middle risk) a more intensive online intervention designed for diverse AMSM engaging in HIV transmission risk behaviors (Keep It Up!), and (3-high risk) the most intensive is a motivational interviewing (MI) intervention that will be delivered by MI therapists via online videochat (Young Men's Health Project).

DETAILED DESCRIPTION:
Adolescent (ages 13-18) men who have sex with men (AMSM) experience a dramatic health disparity as they represent 2% of young people but account for almost 80% of HIV diagnoses in youth. Despite this disproportionate burden, current evidence-based HIV prevention programs focus primarily on adults and heterosexual youth. Because issues affecting sexual health decisions among AMSM are unique, interventions need to be designed to ensure appropriate content that resonates with AMSM. Prevention programs must also be responsive to minority AMSM that experience disparities in incidence or lack of access to prevention services. For example, Hispanics represent 27% of HIV infections among MSM, but Spanish speaking MSM face significant language barriers to accessing HIV services.

Implementation issues are particularly critical as traditional HIV prevention delivery channels have significant limitations for AMSM: few adolescents attend LGBT youth oriented programs, schools place many restrictions on discussions of MSM sexual health, and major questions remain as to the feasibility of enrolling parents of AMSM into HIV prevention programs. With 92% of adolescents (across all races and income levels) going online every day, eHealth interventions represent a critical modality for delivering AMSM- specific intervention material where youth "are." Combining online recruitment with intervention delivery across a range of devices can overcome many access barriers to engagement of AMSM in HIV prevention.

Unfortunately, there will be no single magic solution that will work for all AMSM and public health programmers should not continue to deliver the same fixed intervention when a participant is not responding. Alternatively, stepped-care strategies increase in intensity to meet the needs of those who do not respond to a less intense intervention. Using a Sequential Multiple Assignment Randomized Trial (SMART) design, the investigators will evaluate the impact of a package of increasingly intensive interventions that have already shown evidence of efficacy with diverse adolescent and young adult MSM. The SMART methodology is an ideal approach because SMART designs mimic treatment decisions as they are made in real-world clinical settings, components of traditional RCTs are embedded within the design, and participant data can be used post-hoc to inform decision rules in order to optimize implementation. Collectively the investigators brand this package of eHealth interventions as the SMART Program (Sexual Minority Adolescent Risk Taking). The SMART Program package includes: (1) a universally-delivered, brief, online sexual health education program designed for sexual and gender minority youth regardless of whether they are sexually active ("Queer Sex Ed") (2) a more intensive online intervention designed for diverse AMSM engaging in HIV transmission risk behaviors ("Keep It Up!"); and (3) a more intensive motivational interviewing (MI) intervention that will be delivered by MI therapists via online videochat ("Young Men's Health Project"). The investigators will evaluate the impact of the SMART Program and carefully document implementation context to inform scale out with the following aims:

Aim 1: Evaluate the impact of the SMART Program and its constituent components at reducing HIV risk among AMSM. To do this, the investigators will:

1. Involve diverse AMSM (e.g., Youth Advisory Council) in developmentally adapting existing SMART Program components for AMSM ages 13-18 using the ADAPT-ITT framework.
2. Culturally and linguistically adapt the SMART Program for Spanish speaking Latino AMSM in the US.
3. Embed the SMART Program content into an eHealth platform that will allow access on a range of devices and accommodate updates. Perform alpha and beta testing.
4. Enroll a national sample of 1,938 AMSM who are diverse in terms of race/ethnicity, age, geographic region, socioeconomic status, and sexual experience history.
5. Test the effectiveness of the SMART Program at reducing HIV risk taking behaviors, increasing HIV testing, and improving prevention intentions. Consistent with a SMART design, the investigators operationalize and power the primary test of effectiveness as the first point of randomization, which tests the effectiveness of "Keep It Up!". Additional comparisons will allow the investigators to establish the response rate for "Queer Sex Ed", examine whether the more intensive "Young Men's Health Project" outperforms the less intensive "Keep It Up!" among non-responders to "Queer Sex Ed," and determine whether "Young Men's Health Project" provides added benefit to AMSM who did not respond to "Keep it Up!".

Aim 2: Test if the SMART Program has differential efficacy across important sub-groups of AMSM. Consistent with the RFA, the investigators will test intervention effects within each of the NIH designated health disparity populations (racial/ethnicity minorities, rural, low SES), and by age and language (Spanish).

Aim 3: Evaluate the delivery of the SMART Program nationally to inform scale out and determine cost-effectiveness. To reduce the science-practice gap, the investigators will utilize mixed methods to identify facilitators and barriers to the implementation of the SMART Program using a Hybrid Type 1 Effectiveness-Implementation trial design. The investigators will assess process metrics and indicators of its acceptability among AMSM and key national stakeholders, scale out feasibility, sustainability potential, and conduct a cost analysis to estimate the cost of program implementation compare to monetized benefits.

ELIGIBILITY:
Inclusion Criteria:

* identifying as male-assigned at birth
* reporting attraction to men;
* 13-18 years old
* self-reported HIV-negative at the beginning of the study (or have never been HIV tested/do not know their HIV status)
* able to read English or Spanish,
* has a usable e-mail address, textable phone number, and access to the internet or smart-phone/-device

Exclusion Criteria:

* identifying as female-assigned at birth
* reporting no attraction men
* identifying as under 13 years of age
* identifying as 19 years old or older
* self-reported HIV-positive
* unable to read English or Spanish
* unable to have access to or use email, text messaging, voice calling
* unable to have access to the internet or a smart-phone/-device

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male-assigned at birth
Enrollment: 1306 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Condomless anal sex | 12-months
  Changes in condomless anal sex acts from baseline to 12-months.
Condom Use Intentions Scale | 12-months
  This is a multi-item scale which asks participants about their plans and abilities to use condoms in the future. It has two subscales. The first subscale (Condom Use) asks about participants' likelihood to use condoms with partners. An example item for Condom Use is: "How likely is it that you will use a condom every time you have sex?" The 11-items for this subscale are measured from very unlikely (1) to very likely (4) [averaged min value 1, averaged max value 4]. High values mean a better outcome, or likely condom use with partners. The second subscale (Self-Efficacy) asks participants' ability to use condoms. An example item for Self-Efficacy is: "How confident are you that you would be able to be sure you had condoms with you?" The 5-items for this subscale are measured from not at all confident (1) to extremely confident (7) [averaged min value 1, averaged max value 7]. High values mean a better outcome, or more confidence at using condoms. The two subscales are not combined.
HIV Testing | 12-months
  Participants are asked to self-reported their history of actual getting HIV tested.

SECONDARY OUTCOMES:
HIV Knowledge | Months: 0, 3, 6, 9, 12
  The brief HIV/AIDS Knowledge questionnaire assesses knowledge of transmission and prevention of HIV. Example items that are dichotomously measured as true/false, include: "A person can get HIV by sharing a glass of water with someone who has HIV," "There is a vaccine that can stop people (or adults) from getting HIV," "Using a latex condom or rubber can lower a person's chance of getting HIV," etc.
HIV/AIDS Motivation and Behavioral Skills | Months: 0, 3, 6, 9, 12
  Motivation (e.g. perceived threat of HIV/STI infection, motivation to become safer), social norms (e.g., partners/friends/family members opinions about condom use), and behavioral skills (e.g., negotiating condom use) will be assessed. An example of motivation-based measures would be: "True or False: You really only need to use condoms during one night stands." An example of social norm-based measures would be: "How likely/unlikely is it that you will have sex without a condom because you are afraid of what a partner might do to you if you ask to use condoms?" An example of skills-based measures would be: "How hard would it be for you to discuss safer sex with a partner in a non-sexual setting, such as while riding in your car?" More specific behavioral skills are also measured within the The Health Protective Communication Scale. An example of this would be, "In the past 12 months, have you asked a new sex partner about the number of past sex partners (he/she) had?"
Condom Errors | Months: 0, 3, 6, 9, 12
  An adaptation of the Condom Errors Questionnaire will be asked, which has been found to be predictive of condom breakage and slippage, and STI contraction. An example item from this questionnaire is: "When you used condoms during the LAST 6 MONTHS, how often was the condom package checked for visible damage before having sex?"

OTHER OUTCOMES:
PrEP Knowledge/Experience | Months: 0, 3, 6, 9, 12
  The Knowledge of and Experience with Pre-Exposure Prophylaxis (PrEP) scale (for adolescents) will be used. This is a validated scale that asks questions such as: (Agree/Disagree) "Taking pre-exposure prophylaxis (a pill, also known as PrEP or Truvada) regularly can reduce the risk of contracting HIV from an HIV-positive sex partner."

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mustanski, PhD, Principal Investigator — Northwestern University; Maggie Matson, MPH, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yellin H, Wang Y, Huebner DM, Rodriguez-Diaz CE, Macapagal K, Newcomb ME, Mustanski B, Ruiz MS. An empirical test of the Information-Motivation-Behavioral Skills model of willingness and intention to use HIV pre-exposure prophylaxis among adolescent men who have sex with men. Ann Behav Med. 2025 Jan 4;59(1):kaaf070. doi: 10.1093/abm/kaaf070. PMID 40971723
- [Derived] Mustanski B, Macapagal K, Li DH, Rodriguez-Diaz CE, Saber R, Matson M, Moskowitz DA, Rendina HJ, Laber E, Ryan DT, Newcomb ME. Effectiveness of the smart program: Stepped-care HIV prevention for gay and bisexual adolescent boys. Health Psychol. 2025 Mar;44(3):321-331. doi: 10.1037/hea0001471. PMID 39992778
- [Derived] Sinno J, Macapagal K, Mustanski B. Social Media and Online Dating Safety Practices by Adolescent Sexual and Gender Diverse Men: Mixed-Methods Findings From the SMART Study. J Adolesc Health. 2024 Jan;74(1):113-122. doi: 10.1016/j.jadohealth.2023.07.030. Epub 2023 Oct 4. PMID 37791926
- [Derived] Xavier Hall CD, Wood CV, Hurtado M, Moskowitz DA, Dyar C, Mustanski B. Identifying leaks in the STEM recruitment pipeline among sexual and gender minority US secondary students. PLoS One. 2022 Jun 3;17(6):e0268769. doi: 10.1371/journal.pone.0268769. eCollection 2022. PMID 35658021
- [Derived] Moskowitz DA, Moran KO, Matson M, Alvarado-Avila A, Mustanski B. The PrEP Cascade in a National Cohort of Adolescent Men Who Have Sex With Men. J Acquir Immune Defic Syndr. 2021 Apr 15;86(5):536-543. doi: 10.1097/QAI.0000000000002613. PMID 33399311
- [Derived] Mustanski B, Moskowitz DA, Moran KO, Newcomb ME, Macapagal K, Rodriguez-Diaz C, Rendina HJ, Laber EB, Li DH, Matson M, Talan AJ, Cabral C. Evaluation of a Stepped-Care eHealth HIV Prevention Program for Diverse Adolescent Men Who Have Sex With Men: Protocol for a Hybrid Type 1 Effectiveness Implementation Trial of SMART. JMIR Res Protoc. 2020 Aug 11;9(8):e19701. doi: 10.2196/19701. PMID 32779573
- [Derived] Mustanski B, Moskowitz DA, Moran KO, Rendina HJ, Newcomb ME, Macapagal K. Factors Associated With HIV Testing in Teenage Men Who Have Sex With Men. Pediatrics. 2020 Mar;145(3):e20192322. doi: 10.1542/peds.2019-2322. Epub 2020 Feb 11. PMID 32047100

DOCUMENTS (1):
  • Informed Consent Form (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03511131/ICF_000.pdf